CLINICAL TRIAL: NCT00194714
Title: Phase I/II Study of Combination Immunotherapy for the Generation of HER-2/Neu (HER2) Specific Cytotoxic T Cells (CTL) in Vivo
Brief Title: Vaccine Therapy in Treating Patients With Stage IV HLA-A2 and HER2 Positive Breast or Ovarian Cancer Receiving Trastuzumab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary (Nora) Disis, Professor, University of Washington, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6304; NCI-2016-00895 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 6304 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1000607 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2022-06-21 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: HER2/Neu Positive; HLA-A2 Positive Cells Present; Stage IV Breast Cancer; Stage IV Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (HER-2/neu peptide vaccine) (Experimental): Patients receive HER-2/neu peptide vaccine ID once per month for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: HER-2/neu Peptide Vaccine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: HER-2/neu Peptide Vaccine — Given ID
  Other Names: HER-2-Neu Peptide Vaccine; HER-2/neu Helper-Peptide Vaccine
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects of vaccine therapy and to see how well it works in treating patients with stage IV major histocompatibility complex, class I, A2 antigen (HLA-A2) and human epidermal growth factor receptor 2 (HER2) positive breast or ovarian cancer who are receiving trastuzumab. Giving booster vaccines made from HER2 peptides may help increase HER2 specific immunity and immune memory cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of administering a HER2 cytotoxic T-cell (CTL) peptide-based vaccine (HER-2/neu peptide vaccine) to stage IV breast and ovarian cancer patients receiving maintenance trastuzumab.

II. To quantify and characterize antigen specific T cell subsets specific to HER2 in peripheral blood mononuclear cell (PBMC) of patients after vaccination with a HER2 CTL peptide-based vaccine while receiving maintenance trastuzumab.

SECONDARY OBJECTIVES:

I. To evaluate overall survival (OS) in patients who complete a vaccination series with a HER2 CTL peptide-based vaccine while receiving maintenance trastuzumab.

OUTLINE:

Patients receive HER-2/neu peptide vaccine intradermally (ID) once per month for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1, 3, 6, and 12 months, and then yearly for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have either stage IV breast or ovarian cancer in remission or with stable disease on trastuzumab monotherapy
* HER2 overexpression by immunohistocytochemistry (IHC) of 2+ or 3+, in the primary tumor or metastasis; if overexpression is 2+ by IHC, then patients must have HER2 gene amplification documented by fluorescence in situ hybridization (FISH)
* Subjects must be HLA-A2 positive
* Eligible subjects must have completed appropriate treatment for their primary disease and be off cytotoxic chemotherapy and any immunosuppressive agents such as systemic steroids for at least 30 days prior to enrollment; patients should continue trastuzumab monotherapy throughout the course of this protocol; concurrent hormonal and biphosphonate therapies are allowed
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status score = 0 or 1
* Male subjects must agree to contraceptive use during the study period (7 months) and non-menopausal female subjects must agree to contraception for the remainder of their childbearing years
* Hematocrit >= 30 performed within 60 days of enrollment
* Platelet count >= 100,000 performed within 60 days of enrollment
* White blood cells (WBC) >= 3000/ul performed within 60 days of enrollment
* Stable creatinine =< 2.0 mg/dL or creatinine clearance >= 60 ml/min performed within 60 days of enrollment
* Serum bilirubin < 1.5 mg/dl performed within 60 days of enrollment
* Serum glutamic-oxaloacetic transaminase (SGOT) < 2 x upper limit of normal (ULN) performed within 60 days of enrollment
* Subjects must have recovered from major infections and/or surgical procedures and, in the opinion of the investigator, not have a significant active concurrent medical illness precluding protocol treatment or survival
* Patients must have a baseline left ventricular ejection fraction (LVEF) measured by multi-gated acquisition scan (MUGA) equal to or greater than the lower limit of normal for the radiology facility and if there are two consecutive MUGAS performed while on trastuzumab from the same radiology facility, there cannot be a decrease in LVEF of > 15% from the original MUGA scan

Exclusion Criteria:

* Subjects cannot be simultaneously enrolled on other treatment studies
* Any contraindication to receiving granulocyte-macrophage colony-stimulating factor (GM-CSF) based vaccine products
* Cardiac disease, specifically restrictive cardiomyopathy, unstable angina within the last 6 months prior to enrollment, New York Heart Association functional class III-IV heart failure on active treatment with normalized LVEF on therapy, and symptomatic pericardial effusion
* Active autoimmune disease
* Subjects cannot have an active immunodeficiency disorder, e.g. human immunodeficiency virus (HIV)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05; Primary Completion 2021-03-31 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Disis, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Disis ML, Wallace DR, Gooley TA, Dang Y, Slota M, Lu H, Coveler AL, Childs JS, Higgins DM, Fintak PA, dela Rosa C, Tietje K, Link J, Waisman J, Salazar LG. Concurrent trastuzumab and HER2/neu-specific vaccination in patients with metastatic breast cancer. J Clin Oncol. 2009 Oct 1;27(28):4685-92. doi: 10.1200/JCO.2008.20.6789. Epub 2009 Aug 31. PMID 19720923
- See also: Tumor Vaccine Group, University of Washington — http://depts.washington.edu/tumorvac/
- See also: Fred Hutch - Clinical Trials — http://www.fredhutch.org/en/treatment/clinical-trials.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (HER-2/Neu Peptide Vaccine): Patients receive a HER-2/neu (HER2) specific cytotoxic T cell (CTL) generating peptide vaccine ID once per month for 6 months in the absence of disease progression or unacceptable toxicity. The final dose of peptide vaccine delivered is 1.5 mg (500 mcg/each peptide) admixed with 100 mcg GM-CSF as an adjuvant.
  HER-2/neu Peptide Vaccine: Given ID
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (HER-2/Neu Peptide Vaccine)
Started | 22 (Number of patients consented)
Completed | 21 (Number of patients that received study treatment with the study vaccine)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (HER-2/Neu Peptide Vaccine)
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 49 [33 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Immune Response Measured by IFN-gamma Secreting PBMC Precursor Frequency by ELIspot and HLA-A2 Major Histocompatibility Complex Tetramer Analysis
Description: ELIspot: Increased immune response is defined as spots per well (SPW) greater than 2 standard deviations (SD) above baseline value, remained the same if the mean SPW was within 2 SD of the previous value, or decreased if the mean SPW was greater than 2 SD below the previous value. Two SD is equivalent to a P value of .05 in that there is a 95% probability that the values are statistically significant. T is reported as percentage of patients and their corresponding results.
  HLA-A2 Major Histocompatibility Complex Tetramer Analysis is evaluated using a non-radioactive assay for cell lysis. The HLA-A2 transfected human HER2/neu expressing breast cancer cell line, SKBR3-A2 T cells, expanded after stimulation with immunizing peptide, were added in an effector/target ratio of 40:1. Percent specific lysis was calculated as: ([experimental release-spontaneous releases of cytotoxic T-lymphocyte cells and target cells]/[maximum release-spontaneous release of target cells])X100.
Time Frame: Up to 1.5 years (12 months following the last vaccination)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (HER-2/Neu Peptide Vaccine)
Number analyzed (Participants) | 19
Participants
  HLA-A2 Results: Significantly augmented immune response | 14
  HLA-A2 Results: Did not have augmentation of immune response | 4
  HLA-A2 Results: Decrease in immune response | 1
  ELIspot: Significantly augmented immune response | 16
  ELIspot: Did not have augmentation of immune response | 3
  ELIspot: Decrease in immune response | 0

2. Primary Outcome: Number of Adverse Events Graded Using National Cancer Institute (NCI) Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0
Description: Descriptive statistics will be used to summarize changes from baseline. At the point the participant signs consent and before they start vaccine we record their existing baseline events (symptoms and diagnoses) and assign a grade to them (see below). Once a participant starts vaccine treatment adverse event AEs were recorded if they are new to the participant or if they increased in severity over their baseline.
  Grade refers to the severity of the AE. The CTCAE v3.0 displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: Up to 7 months (30 days following the last vaccination)
Population: We recorded a total of 573 individual adverse events from baseline through follow-up evaluation for 21 patients. The data below represents the total number of events by Grade using Common Terminology Criteria for Adverse Events v3.0 (CTCAE)
Measure: Number; unit: adverse events
Arm/Group | Treatment (HER-2/Neu Peptide Vaccine)
Number analyzed (Participants) | 21
adverse events
  Grade 1 | 508
  Grade 2 | 60
  Grade 3 | 4
  Grade 4 | 1

3. Secondary Outcome: Overall Survival
Description: Survival for the Stage IV breast cancer patients will be compared to historical control.
Time Frame: Up to 5 years
Population: These are interim results: We are still monitoring overall survival.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (HER-2/Neu Peptide Vaccine)
Number analyzed (Participants) | 21
Participants
  Alive | 10
  Deceased | 11

ADVERSE EVENTS:
Time Frame: Patients were evaluated during the study treatment (6 months) and then for 5 additional years after that where we were evaluating any potential development of long-term autoimmune disease.
Description: We used CTCAE v3.0 for this study. The adverse events reported here include all events regardless of whether they were unrelated and related to study treatment). Please note that these tables record every adverse event for every subject regardless of severity. For example, a subject may have an injection site reaction at each of the three vaccines where another may not. Each one of these injection site reactions is recorded for that one subject.
Arm/Group | Treatment (HER-2/Neu Peptide Vaccine)
All-Cause Mortality (participants affected / at risk) | 11/21
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (HER-2/Neu Peptide Vaccine) (N=21)
CNS Cerebrovascular Ischema (Nervous system disorders) | 1 (1) — This was a Grade 4 event that was unrelated to the study treatment
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) — This was a Grade 2 event that was determined to be possibly related to the study treatment
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) — This was recorded as a Grade 3 event that was possibly related to the study treatment. This occurred after the patient spent time in the sun.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (HER-2/Neu Peptide Vaccine) (N=21)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Not related to study treatment
Lymphopenia (Investigations) | 10 (33) — 28 events were deemed related; 5 were deemed unrelated to the study treatment
Anemia (Investigations) | 9 (11) — 4 events were deemed related; 7 events were deemed unrelated to study treatment
Platelets low (Investigations) | 3 (6) — 4 events were deemed related; 2 events were deemed unrelated to the study treatment
Leukopenia (Investigations) | 10 (29) — 27 events were deemed related; 2 were deemed unrelated to study treatment
Leukocytosis (Investigations) | 1 (1) — Due to steroids; Unrelated to study treatment
Eosinophilia (Investigations) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 7 (9)
Palpatations (Cardiac disorders) | 6 (9) — 2 of the events were deemed related; 7 of the events were deemed unrelated to study treatment
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1) — This event was deemed possibly related to study treatment
Hypertension (Vascular disorders) | 4 (5) — Not related to study treatment
Left ventricular systolic dysfunction (Cardiac disorders) | 3 (3) — Events deemed related to study treatment
Chest tightness (Cardiac disorders) | 1 (1) — Not related to study treatment
Fever (General disorders) | 4 (4) — 2 events were deemed related; 2 events were deemed unrelated to study treatment
Rigors/Chills (General disorders) | 12 (20) — 16 events were deemed related; 4 events were deemed unrelated to study treatment
Fatigue (General disorders) | 20 (43) — 38 events were deemed related; 4 events were deemed unrelated
Sweating (General disorders) | 1 (1)
Weepiness (General disorders) | 1 (1) — Not related to study treatment
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Injection Site Reaction (General disorders) | 20 (68) — All events were related to administration of study treatment
Flushing (Vascular disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Pruritis/Itching (Skin and subcutaneous tissue disorders) | 12 (22) — 20 events deemed related; 2 events deemed unrelated to study treatment
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 (8)
Rash/acneiiform (Skin and subcutaneous tissue disorders) | 4 (7)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 4 (5) — Events are related to study treatment
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2) — Not related to study treatment
Alopecia (Skin and subcutaneous tissue disorders) | 3 (5) — 3 events deemed related; 2 events deemed unrelated to study treatment
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) — Not related to study treatment
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) — Related to study treatment
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) — Related to study treatment
Hot flashes (Vascular disorders) | 2 (2) — 1 event was related; 1 event was not related to study treatment
Diarrhea (Gastrointestinal disorders) | 11 (17) — 6 events are deemed related; 11 events are deemed unrelated to study treatment
Nausea (Gastrointestinal disorders) | 12 (22) — 13 events deemed related; 9 events deemed unrelated to study treatment
Vomiting (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (4) — Not related to study treatment
Mucositis/stomatisis (functional/symptomatic) (Gastrointestinal disorders) | 1 (1) — Not related to study treatment
Blood in stool (Gastrointestinal disorders) | 1 (2) — Not related to study treatment
Hemorrhage, GU (Gastrointestinal disorders) | 1 (1)
Infection with normal ANC or GRA1 or 2 neutrophils (Infections and infestations) | 10 (11) — Not related to study treatment
Infection without neutrophils (Infections and infestations) | 1 (1) — Not related to study treatment
Edema:limb (General disorders) | 8 (16) — 8 events were deemed related; 8 events were deemed unrelated to study treatment
Edema: Head and neck (General disorders) | 1 (1)
Swelling left breast (Reproductive system and breast disorders) | 1 (1) — Not related to study treatment
Lymphnode pain (Blood and lymphatic system disorders) | 1 (1)
aspartate aminotransferase (AST)/SGOT (Investigations) | 2 (6) — 1 event deemed related; 5 events deemed unrelated to study treatment
Hypokalemia (Metabolism and nutrition disorders) | 2 (6) — Not related to study treatment
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) — Not related to study treatment
Alanine aminotransferase increased (ALT)/SGPT (Metabolism and nutrition disorders) | 2 (6) — Not related to study treatment
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) — Not related to study treatment
Creatinine (Investigations) | 3 (8) — 1 event was related; 7 events unrelated to study treatment
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3) — Not related to study treatment
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to study treatment
Dizziness (Nervous system disorders) | 8 (11) — 8 events deemed related; 3 events deemed unrelated to study treatment
Confusion (Psychiatric disorders) | 1 (1) — Not related to study treatment
Neuropathy: sensory (Nervous system disorders) | 3 (4)
Neuropathy: motor (Nervous system disorders) | 2 (3) — Not related to study treatment
Syncope (Nervous system disorders) | 1 (1)
Pain - Headache (Nervous system disorders) | 14 (42) — 27/42 events were deemed related to the study treatment
Pain - Abdomen NOS (Gastrointestinal disorders) | 4 (7)
Pain - Leg cramps (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Back (Musculoskeletal and connective tissue disorders) | 4 (7)
Pain - Arlthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Chest Wall (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Rib (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Injection site (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain - Breast (Reproductive system and breast disorders) | 1 (1)
Pain - Lung (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pain - Lymphnode (Blood and lymphatic system disorders) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (43) — 33 events were deemed related; 10 events were deemed unrelated to study treatment
Pain - Pleuritic (Respiratory, thoracic and mediastinal disorders) | 1 (1) — After liver biopsy
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (6) — Not related to study treatment
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hemorrhage/Bleeding associated with surgery, intra-operative or postoperative (Surgical and medical procedures) | 1 (1) — Not related to study treatment
Urine leukocytes (Renal and urinary disorders) | 1 (2) — Not related to study treatment
Flu-like syndrome (General disorders) | 7 (10) — Related to study treatment
Vision - blurred (Eye disorders) | 1 (1) — Not related to study treatment
Hypotension (Cardiac disorders) | 1 (1) — This event was Grade 2 and deemed related to the study treatment
Infection Other - PAC infection (Infections and infestations) | 1 (1) — This was a Grade 2 events that was unrelated to the study treatment
Infection Other - Cold (Infections and infestations) | 1 (1) — Unrelated to study treatment
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) — Unrelated to study treatment
Pain - Extremity Limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dry Eye Syndrome (Eye disorders) | 1 (1) — This event was deemed unrelated to study treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-04-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT00194714/Prot_SAP_000.pdf
  • Informed Consent Form (2016-04-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT00194714/ICF_001.pdf